CLINICAL TRIAL: NCT00696540
Title: Safety and Efficacy of Hypertonic Vrs. Normal Saline as Diluent of Salbutamol to Reduce Respiratory Distress in Outpatients With the Clinical Diagnosis of Bronchiolitis During the RSV Epidemic.
Brief Title: Hypertonic Saline for Outpatient Bronchiolitis
Acronym: Hypertonic
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Diego Portales (Other)
Collaborators: Clínica Vespucio, Santiago, Chile (Unknown)
Responsible Party: Irmeli Roine, Facultad de Ciencias de la Salud, Universidad Diego Portales, Santiago. Chile
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UDP-CT1-08
Record Dates: First submitted 2008-06-09; First posted 2008-06-12 (Estimated); Last update posted 2008-06-12 (Estimated); Status verified 2008-06

CONDITIONS: Bronchiolitis; Respiratory Distress
Keywords: Bronchiolitis, respiratory distress, hypertonic saline
MeSH Terms: conditions — Bronchiolitis; Dyspnea | interventions — Saline Solution, Hypertonic; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Salbutamol is diluted in hypertonic (3%) saline.
  Interventions: Drug: Inhalation of salbutamol diluted in hypertonic saline
- 2 (Active Comparator): Salbutamol is diluted in normal (0.9%) saline.
  Interventions: Drug: Inhalation of salbutamol diluted in normal saline

INTERVENTIONS:
Drug: Inhalation of salbutamol diluted in hypertonic saline — The first of 3 nebulizations of 0.5 mg of Salbutamol is diluted in 3.5 ml of hypertonic (3%) saline. The second and the third are diluted in normal (0.9%) saline.
  Other Names: Albuterol diluted in hypertonic saline
  Arms: 1
Drug: Inhalation of salbutamol diluted in normal saline — The 3 nebulizations of 0.5 mg of Salbutamol are diluted in 3.5 ml of normal (0.9%) saline.
  Other Names: Albuterol diluted in normal saline
  Arms: 2

SUMMARY:
We will study if small children who become ill with respiratory distress during the RSV epidemic are better relieved with salbutamol nebulizations diluted in hypertonic (3%), instead of normal (0.9%) saline.

DETAILED DESCRIPTION:
In Santiago, Chile, a near collapse of health services is a notorious feature of every winter when vast numbers of small children line for attention because of respiratory distress caused by a probable RSV infection.

Our study will examine if nebulized salbutamol diluted in hypertonic (3%), instead of normal (0.9%) saline, provides better relief in outpatients.

If hypertonic saline proves safe and effective, the patients could be better managed and the pressure for attention diminished at a low cost, by a simple change in the saline ampule.

ELIGIBILITY:
Inclusion Criteria:

1. Age 1 to 24 months
2. Mild to moderate respiratory distress (Tal score below 9)
3. Up to 5 days of respiratory symptoms, including today
4. Expiratory wheezing heard on chest auscultation
5. Indication of salbutamol nebulization treatment by attending physician

Exclusion Criteria:

1. Two prior episodes of wheezing
2. Premature birth (below 38 weeks), if below 6 months of age
3. Lobar pneumonia
4. Body temperature above 38 degree Celsius
5. Use of salbutamol during the previous 6 hours
6. Pulse oxymetry reading below 90%
7. Congenital heart disease
8. Chronic pulmonary disease: Asthma, cystic fibrosis, bronchopulmonary dysplasia
9. Other chronic or genetic condition or disease

Ages: 1 Month to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 74 (Estimated)
Dates: Start 2008-06; Primary Completion 2008-09 (Estimated); Study Completion 2008-10 (Estimated)

PRIMARY OUTCOMES:
Change in the respiratory distress score (Tal) between the basal score and the final score after 3 salbutamol nebulizations | 1 hour

SECONDARY OUTCOMES:
Change in the respiratory distress score (Tal) between the basal score and the first nebulization | 15 to 20 minutes
Change in the respiratory distress score (Tal) between the basal score and the second nebulization | 15 to 20 minutes after the first nebulization
Change in pulse oxymetry reading between the basal score and after each of the three nebulizations | 1 hour
Change in cardiac frequency, irritability, general condition or anything else between the basal score and the first, second and third nebulization | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Irmeli Roine, MD, PhD, Principal Investigator — University Diego Portales; Ricardo Mercado, MD, Study Director — Clinica Vespucio, Santiago, Chile
Locations (1):
- Clínica Vespucio, Santiago, Chile

REFERENCES:
- [Background] Sarrell EM, Tal G, Witzling M, Someck E, Houri S, Cohen HA, Mandelberg A. Nebulized 3% hypertonic saline solution treatment in ambulatory children with viral bronchiolitis decreases symptoms. Chest. 2002 Dec;122(6):2015-20. doi: 10.1378/chest.122.6.2015. PMID 12475841
- [Background] Mandelberg A, Tal G, Witzling M, Someck E, Houri S, Balin A, Priel IE. Nebulized 3% hypertonic saline solution treatment in hospitalized infants with viral bronchiolitis. Chest. 2003 Feb;123(2):481-7. doi: 10.1378/chest.123.2.481. PMID 12576370